CLINICAL TRIAL: NCT06330077
Title: A Phase 2 Trial Assessing Ifenprodil as a ReMyelinating repurpOsed Drug in Multiple Sclerosis
Brief Title: Ifenprodil as a ReMyelinating repurpOsed Drug in Multiple Sclerosis
Acronym: MODIF-MS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP200027; 2021-003584-99 (EudraCT Number)
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis; Remitting Relapsing Multiple Sclerosis
Keywords: Multiple Sclerosis; Ifenprofil; Combination of magnetic resonance imaging (MRI) and positron emission tomography (PET); 18f-Florbetaben; Remyelination
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — ifenprodil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ifenprodil (Experimental): Ifenprodil : 20mg three time a day (60mg/day). Patients will have an escalation of dose over 48 hours (from Day 1) in order to achieve at the end of the 144 hours (6 days, Day 6) a dose of 60mg/day.
  Interventions: Drug: Ifenprodil
- Placebo (Placebo Comparator): Placebo of ifenprodil : 20mg three time a day (60mg/day). Patients will have an escalation of dose over 48 hours (from Day 1) in order to achieve at the end of the 144 hours (6 days, Day 6) a dose of 60mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifenprodil — Treatment administration
  Arms: Ifenprodil
Drug: Placebo — Treatment administration
  Arms: Placebo

SUMMARY:
Multiple sclerosis (MS) is the most frequently acquired demyelinating disease and the first cause of non-traumatic chronic disability in young adults. Major progress has been achieved in the treatment of MS through the development of therapies targeting the adaptative immune system, which drastically reduce the relapse rate, with various efficiency and safety profiles (Ontaneda, 2015). However, these drugs generally fail to prevent disability worsening along the disease course, and we are now assisting to a shift in therapeutic objectives from the development of new immune drugs towards the identification of therapeutic strategies that could prevent neurodegeneration by promoting myelin regeneration (Stangel, 2017; Stankoff, 2016), in order to prevent neurological disability in MS (Irvine and Blakemore, 2008; Patrikios, 2006; Duncan I, 2017, Bodini, 2016).

Among the first candidate compounds developed to promote remyelination was the anti Lingo1 antibody, which enhance remyelination (Mi, 2009). Medium and large throughput screening of drug libraries subsequently identified several chemical classes of compounds with strong promyelinating properties, such as the antifongic drug miconazole (Najm, 2015) or the muscarinic antagonist clemastine (Wei, 2014). A recent innovative trial has investigated the effect of clemastine, compared to placebo, in a small sample of subjects (25 patients per group) and showed that clemastine could significantly improve the optic nerve conduction speed which reflecting myelin integrity and functionality (Green, 2017).

Our preclinical research has allowed us to identify ifenprodil as a powerful drug to promote myelin repair in vitro and in vivo across species. In parallel our team recently pioneered and optimized a PET imaging approach for quantifying remyelination in the whole brain, that allowed to enhance the sensitivity to detect the myelin repair process, and showed that patients are characterized by heterogeneous profiles of spontaneous remyelination profiles that are closely linked to disability accrual (Bodini, 2016).

ELIGIBILITY:
Inclusion Criteria:

-

Patients:

1. Signed informed consent form at pre-inclusion visit
2. Age between 18 years and 55 years, inclusive, at time of pre-inclusion visit.
3. Patient with a RR form of MS according McDonald criteria 2017 at pre-inclusion visit
4. Able to comply with the study protocol and to understand the purpose and risks of the study, in the investigator's judgment
5. Social security registration (AME excluded) at time of pre-inclusion visit
6. At least one eye with a P100 latency > 118ms on visual evoked potential at baseline (defining the qualifying eye) at time of pre-inclusion visit
7. Retinal nerve fibre layer thickness on spectral-domain optical coherence tomography [OCT] > 70 μm in the VEP qualifying eye (to increase the likelihood that the number of surviving axons is sufficient to provide the substrate for remyelination to occur) at time of pre-inclusion visit
8. Patient under disease modifying therapy (first or second line approved immune active therapy) or patient without any DMT at time of pre-inclusion visit
9. EDSS score ≤ 6 at time of pre-inclusion visit
10. For women of childbearing potential : Efficient contraception include oral contraception, intrauterine devices hormonal device, intrauterine hormone-releasing system, sterilization method and other forms of contraception with failure rate <1%)

    * Healthy Volunteers

1. Signed informed consent form 2. Age between 18 years and 55 years, inclusive 3. All female subjects of childbearing potential must practice effective contraception include oral contraception, intrauterine devices hormonal device, intrauterine hormone-releasing system, sterilization method and other forms of contraception with failure rate <1%) 4. Able to comply with the study protocol, in the investigator's judgment 5. Social security registration (AME excluded)

Exclusion Criteria:

Patients

1. Patient with an acute NORB in the last 6 months prior to pre-inclusion visit
2. Patient with a clinical relapse other than NORB in the last 6 months prior to pre-inclusion visit
3. Patients having received methylprednisolone infusion in the last 4 weeks prior to pre-inclusion visit
4. Contraindications to investigational medicinal products (ifenprodil/placebo) and to auxiliary medicinal products (gadolinium, [18F]-florbetaben)
5. Inability to complete an MRI (contraindications for MRI include but are not restricted to weight ≥ 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, contraindication to gadoteric acid etc.).
6. PET imaging performed in the past 12 months as part of clinical research
7. History or incidental discovery of significant cardiac conduction block
8. Orthostatic hypotension Syndrome define as a drop of > 20 mmHg in systolic, and/or > 10 mmHg in diastolic between lying down and immediate standing
9. Known long QT syndrome or long QT syndrome (the limit is defined at 450 ms on corrected QT) highlighted during the pre-inclusion visit
10. Any uncontrolled general (cancer, infectious, hematologic, hepatic, immunologic, endocrinologic, neurologic, dermatologic, psychiatric, allergic, renal, or cardiovascular) disease.
11. Creatinine clearance < 60 ml/min at pre-inclusion visit
12. ASAT, ALAT of alkaline phosphatase > 3-fold the upper limit normal at pre-inclusion visit
13. Know Galactosemia, glucose malabsorption or lactase deficiency
14. Known of lack of peripheral venous access or lack of peripheral venous access highlighted during the pre-inclusion visit
15. Thrombocytopenia with platelets < 100 000/mm3
16. Pregnancy and/or lactating women
17. Legal protection (curatorship or tutorship)
18. Deprive of freedom or under security measure
19. Participation in another interventional trial evaluating a health product or any randomized trial or being in the exclusion period at the end of a previous study
20. Refusal to be informed in case of clinically significant incidental discovery after MRI
21. Patient treated for hypertension with the following drugs blocking the alpha-adrenergic system either in periphery (prazosine, urapidil, moxisylyte, labetalol) or centrally (clonidine, monoxidine, methyldopa)

Healthy Volunteers

1. Inability to complete an MRI (contraindications for MRI include but are not restricted to weight ≥ 140 kg, pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, etc).
2. Impossibility to complete a PET scan: pregnancy, nuclear medicine irradiation for clinical research in the year preceding baseline visit.
3. Contraindication to auxiliary medicinal products ([18F]-florbetaben)
4. Known presence of any neurological disorders
5. Pregnancy and/or lactation
6. Lack of peripheral venous access
7. Terminal renal insufficiency (Creatinin clearance < 60 ml/min)
8. Legal protection (curatorship or tutorship)
9. Deprive of freedom or under security measure
10. Participation in another interventional trial evaluating a health product or any randomized trial or being in the exclusion period at the end of a previous study
11. Refusal to be informed in case of clinically significant incidental discovery after MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in P100 latency according to visual evoked potential. | Between months 6 and months 12
  Assess the efficacy of ifenprodil on the remyelination of the optic nerve measured as the improvement of P100 latency, assessed using full field visual evoked potentials.

SECONDARY OUTCOMES:
Proportion of voxels within white matter lesions classified as remyelinating | Between 6 months and 12 months
  Change in remyelination potential measured by PET-MR Between M6 (end of run-in, calculation of pre-treatment remyelination potential, randomization) and M12 (end of follow-up, calculation of post-treatment remyelination potential) in each group.
Proportion of remyelinating voxels extracted in cortical regions from magnetization transfer imaging (MTR) acquisitions | Between 6 months and 12 months
  Change in the proportion of remyelinating voxels extracted in cortical regions from MTR acquisitions (as cortical myelin in not assessed by PET) between M6 and M12 in each group
Change in amplitude of P100 on to visual evoked potential | Between 6 months and 12 months
  o determine whether the treatment by ifenprodil could influence axonal damage in the visual pathway assessed by the amplitude of P100
Change in retinal nerve fibre layer (RNFL) and ganglion cell complex (GCC) thickness on OCT | Between 6 months and 12 months
  To determine whether the treatment by ifenprodil could influence neurodegeneration measured by optical coherence tomography (OCT) parameters in each group
Change in blood concentration of NfL fragments | From Pre-inclusion visit to 6 months and from 6 months to 9 months and 6 months to 12 months
  To determine whether the treatment by ifenprodil could influence axonal damage assessed by the blood concentration of neurofilament light chain (NfL) in each group
Change in the brain atrophy rate | From baseline to 6 months and 6 months to 12 months
  To determine whether the treatment by ifenprodil could influence white matter lesions load or brain atrophy rate in each group
The correlation between the change in the proportion of remyelinating voxels extracted in white matter lesions from [18F]florbetaben PET acquisitions | Between 6 months and 12 months and the pre-treatment individual remyelination profiles as determined during the Run-in period
  To determine whether the efficacy of ifenprodil is influenced by endogenous remyelination profiles assessed in the run-in period, and to describe the profile of optimal responders
The comparison of the proportion of remyelinating voxels extracted in white matter lesions from [18F]florbetaben PET acquisitions | Between 6 months and 12 months
  To assess whether the disease modifying therapies received during the study influence the remyelination level and/or the ifenprodil effect on remyelination
Incidence of adverse drug reactions | Between inclusion and 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Neurologique Pierre WERTHEIMER - HCL, Bron
  - Groupe Hospitalier Pitié Salpêtrière - APHP, Paris

IPD SHARING:
Plan to Share IPD: Undecided